CLINICAL TRIAL: NCT00156884
Title: A Randomized Phase II Trial of Strontium-89 With or Without Cisplatin for the Palliation of Bone Pain Secondary to Hormone Refractory Prostate Cancer
Brief Title: A Trial of Strontium +/- Cisplatin for the Palliation of Bone Pain Secondary to Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alberta Health services (Other)
Collaborators: The Prostate Cancer Research Foundation of Canada (Other); Amersham Health (Industry)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUPPS2
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2008-08

CONDITIONS: Hormone Refractory Prostate Cancer; Bone Metastases
Keywords: prostate cancer; cisplatin; strontium-89; phase II
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Strontium-89; Cisplatin

INTERVENTIONS:
Drug: strontium-89
Drug: cisplatin

SUMMARY:
This study is designed to determine whether the combination of low dose cisplatin and strontium-89 shows clinical promise for the symptomatic treatment of bone metastases in hormone refractory prostate cancer.

DETAILED DESCRIPTION:
This study is designed to determine whether the combination of low dose cisplatin and strontium-89 shows clinical promise for the symptomatic treatment of bone metastases in hormone refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the prostate
* life expectancy > 3 months,
* symptomatic from bone metastases
* radiologic evidence of metastatic bone disease
* stable level of pain control
* >18 years
* ability to complete assessments
* prior treatment (chemo) > 4 weeks previous
* discontinued anti-androgens for > 4 weeks

Exclusion Criteria:

* prior strontium therapy
* previous hemibody RT within 6 weeks
* previous cytotoxic chemotherapy within 4 weeks
* use of bisphosphonate medications within 4 weeks
* change in steroid dose within 4 weeks
* active uncontrolled infection
* impending or present spinal cord compression
* significant neurological disorder
* impending pathological fracture
* severe urinary incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2003-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Palliative pain response
analgesic response

CONTACTS AND LOCATIONS:
Overall Officials: Bernie Eigl, MD, Principal Investigator — Alberta Cancerboard; Jackson Wu, Principal Investigator — Alberta Cancerboard
Locations (2):
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Agency, Vancouver, British Columbia